CLINICAL TRIAL: NCT02797015
Title: A Phase I, Multicenter, Randomized, 12-Week, Open-Label Study to Evaluate the Multiple Dose Pharmacokinetics and Pharmacodynamics of RPC 1063 in Patients With Relapsing Multiple Sclerosis
Brief Title: Pharmacokinetics and Pharmacodynamics Study of RPC1063 in RMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RPC01-1001
Record Dates: First submitted 2016-05-26; First posted 2016-06-13 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Multiple Sclerosis
Keywords: MS; RMS; Multiple Sclerosis; Relapsing Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 mg RPC1063 (Experimental): 1 mg RPC1063 oral capsule daily
  Interventions: Drug: RPC1063
- 0.5 mg RPC1063 (Experimental): 0.5 mg RPC1063 oral capsule daily
  Interventions: Drug: RPC1063

INTERVENTIONS:
Drug: RPC1063 — Oral capsule daily

SUMMARY:
The purpose of this study is to learn about the pharmacokinetics and pharmacodynamics of RPC1063 in RMS.

DETAILED DESCRIPTION:
The purpose of this study is to characterize the full pharmacokinetic and pharmacodynamics profiles of RPC1063 in patients with relapsing multiple sclerosis (RMS) following multiple-dose administration of the two different dosing regimens that are being evaluated in the Phase 3 RMS studies.

ELIGIBILITY:
Key Inclusion Criteria:

* MS, as diagnosed by the revised 2010 McDonald criteria
* Exhibits a relapsing clinical course consistent with RMS and history of brain MRI lesions consistent with MS
* Expanded disability status scale (EDSS) score between 0 and 6.0

Key Exclusion Criteria:

* Primary progressive MS
* Clinically relevant cardiovascular conditions or other relevant diseases that could impact the implementation or interpretation of the trial, or put the patient at risk

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 24 hours after the last RPC1063 dose on Day 85
  Maximum plasma concentration (Cmax)
Area under the plasma concentration-time curve (AUC) | Approximately 3 months
  Area under the plasma concentration-time curve (AUC)

SECONDARY OUTCOMES:
Adverse Events | Up to 28 days after the last RPC1063 dose
  Number of participants with treatment-emergent adverse events
EDSS (Expanded Disability Status Scale) | Up to the last RPC1036 dose on Day 85
  Changes from baseline in EDSS
Pharmacodynamic response measured in change from baseline in Absolute Lymphocyte Count | Up to 28 days after the last RPC1063 dose
  Pharmacodynamic response measured in change from baseline in Absolute Lymphocyte Count (absolute and %)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Breastlink Medical Group, Inc., Long Beach, California
  - Multiple Sclerosis Center at UCSF, San Francisco, California
  - Raleigh Neurology Associates PA, Raleigh, North Carolina
  - Neurology and Neuroscience Associates Inc., Akron, Ohio
  - Hope Neurology MS Center, Knoxville, Tennessee
  - Central Texas Neurology Consultants PA, Round Rock, Texas

REFERENCES:
- [Derived] Harris S, Tran JQ, Southworth H, Spencer CM, Cree BAC, Zamvil SS. Effect of the sphingosine-1-phosphate receptor modulator ozanimod on leukocyte subtypes in relapsing MS. Neurol Neuroimmunol Neuroinflamm. 2020 Jul 31;7(5):e839. doi: 10.1212/NXI.0000000000000839. Print 2020 Sep. PMID 32737072